CLINICAL TRIAL: NCT02179905
Title: Brain Imaging, Heart Rate Variability and Serum Fatty Acid in Subjects With Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKH-8302-102-DR-14
Record Dates: First submitted 2014-06-04; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: MRI; Heart rate variability; Fatty acid
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Irritable bowel syndrome, Control

SUMMARY:
This study is to analyze the relationship between brain structure, the heart rate variability and the serum fatty acid component of the irritable bowel syndrome patients.

DETAILED DESCRIPTION:
Several studies showed that the gray matter and white matter of the brain related to the symptoms of irritable bowel syndrome patients.

The investigators study is to analyse the relationship between thickness of cortex of irritable patients, the sympathetic tone and the serum fatty acid component of the irritable bowel syndrome patients. It is to clarify the mechanism of irritable bowel syndrome, whether the symptoms of irritable bowel syndrome are related to the thickness of cortex or inflammation status of the body.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 20 and 50 years old
* meet Rome III criteria

Exclusion Criteria:

* colon and small intestinal disease
* psychiatric disease patients
* patients received major surgery in the past 5 years
* diabetic patients
* patients with metal implant

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Irritable bowel syndrome patients, Control
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The relationship between brain structure, heart rate variability and fatty acid of the irritable bowel syndrome patients. | Patients who suffered from IBS for more than 5 years.

SECONDARY OUTCOMES:
The relationship between thickness of brain cortex and the symptoms of irritable bowel syndrome | Patients who suffered from IBS for more than 5 years.

OTHER OUTCOMES:
The relationship between heart rate variability and symptoms of irritable bowel syndrome patients. | Patients who suffered from IBS for more than 5 years.
The relationship between component of fatty acid and symptoms of irritable bowel syndrome patients. | Patients who suffered from IBS for more than 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan